CLINICAL TRIAL: NCT06962891
Title: Validation of a Proteomic Biomarker to Predict Progression of Chronic Kidney Disease
Acronym: KidneySign
Status: Active, not recruiting | Type: Observational
Sponsor: Angel Argiles (Industry)
Collaborators: Medical University Innsbruck (Other); Klinikum Bayreuth GmbH (Industry); University of Skövde (Other); RWTH Aachen University (Other); RD Néphrologie SAS (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Paul Sabatier of Toulouse (Other)
Responsible Party: Sponsor-Investigator, Angel Argiles, Dr, RD Néphrologie SAS
Organization: RD Néphrologie SAS (Industry)
Other Study IDs: KidneySign Prospective Study; 20230529-3204 (Registry Identifier: Studienregister des LKH - Universitätskliniken Innsbruck); 2024-A00107-40 (Other: ANSM ID-RCB)
Record Dates: First submitted 2025-04-30; First posted 2025-05-08 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease(CKD); Progression, Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma, serum, spot urine, 24-hour collection urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CKD patients: adults with eGFR between 25 and 65 mL/min/1.73m²
  Interventions: Diagnostic Test: CKD progression biomarker

INTERVENTIONS:
Diagnostic Test: CKD progression biomarker — We will evaluate the CKD progression biomarker at baseline and evaluate 1-year CKD progression afterwards.

SUMMARY:
The goal of this longitudinal observational study is to estimate the performances of a candidate proteomic biomarker to identify patients at short term risk of chronic kidney disease (CKD) progression, in CKD patients attending nephrology visits in 3 participating centres. The primary endpoint of CKD progression is defined as a relative change in eGFR observed at 1 year below -10%. The performance of the candidate biomarker will be compared to performances of UAE and KFRE equations.

Participants will attend two study visits (baseline and 1-year), with clinical evaluation including kidney parameters (eGFR, urinary albumin excretion (UAE)) and collection of biological samples (plasma, serum, urine) for candidate proteomic biomarker evaluation. If planned in routine, patients will also have creatinine clearance estimation from 24-hour urine collection, kidney echography and kidney biopsy, sample biobanking and/or questionnaires and interviews on social and ethical aspects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients
* over 18 years and below 85 years of age at recruitment
* Chronic kidney disease (CKD)
* eGFR of 25-65 mL/min/1.73m2 (CKD-EPI formula)
* Beneficiary of health insurance
* Must be able to communicate with the investigator
* Written informed consent must be provided before participation.

Exclusion Criteria:

* History of renal transplantation
* Current episode of Acute Kidney Injury
* Any clinically significant disorder, which in the Investigator's opinion could interfere with the results of the trial.
* Known or suspected abuse of alcohol or narcotics
* Current pregnancy
* Inability to give written informed consent
* Protected adults

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CKD patients attending nephrology medical visits
Sampling Method: Non-Probability Sample
Enrollment: 213 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Relative eGFR change | 1 year
  Difference in eGFR after 1-year divided by baseline eGFR estimated with CKD-EPI formula

SECONDARY OUTCOMES:
Major Adverse Renal Events (MARE) | 1 year
  Composite endpoint defined by the occurrence of any of the following: worsening of kidney disease (-40% eGFR, doubling of creatinine), ESKD (dialysis therapy or renal transplantation), death of any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Angel Argiles, Principal Investigator — RD Néphrologie, Néphrologie Dialyse St Guilhem
Locations (3):
- Medizinische Universität Innsbruck, Innsbruck, Austria
- Néphrologie Dialyse St Guilhem, Sète, France
- Klinikum Bayreuth GmbH, Bayreuth, Germany

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- See also: Project website — https://kidneysign.eu/